CLINICAL TRIAL: NCT06853769
Title: A Prospective, Single-arm, Single-center Exploratory Clinical Study of Anlotinib in Combination With Penpulimab and Conventional Chemoradiotherapy for the Neoadjuvant Treatment of Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Therapy for Locally Advanced Rectal Cancer
Acronym: LARC-nCR01
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-563
Record Dates: First submitted 2024-09-11; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — penpulimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Penpulimab 200mg IV D1 Anlotinib 12mg P.O. QD D1-14 Radiation therapy 1.8-2Gy/50-55Gy
  Chemotherapy:
  Capecitabine 800mg/m2 P.O. BID D1-D14, or capecitabine plus oxaliplatin 130mg/m2. Every 21 days is 1 cycle In the above regimen, two cycles of targeted therapy (chemotherapy + immunotherapy + targeted therapy) are synchronized during radiotherapy; After the end of radiotherapy, two cycles of adjuvant chemo-immunotherapy (chemotherapy + immunotherapy) were continued.
  Interventions: Drug: Anlotinib hydrochloride,Penpulimab

INTERVENTIONS:
Drug: Anlotinib hydrochloride,Penpulimab — Penpulimab 200mg IV D1 Anlotinib 12mg P.O. QD D1-14
  Other Names: FOCUS

SUMMARY:
This study aims to evaluate the clinical efficacy and safety of anlotinib in combination with penpulimab and conventional chemoradiotherapy for the neoadjuvant treatment of locally advanced rectal cancer

DETAILED DESCRIPTION:
Penpulimab 200mg IV D1 Anlotinib 12mg P.O. QD D1-14 Radiation therapy 1.8-2Gy/50-55Gy

Chemotherapy:

Capecitabine 800mg/m2 P.O. BID D1-D14, or capecitabine plus oxaliplatin 130mg/m2. Every 21 days is 1 cycle In the above regimen, two cycles of targeted therapy (chemotherapy + immunotherapy + targeted therapy) are synchronized during radiotherapy; After the end of radiotherapy, two cycles of adjuvant chemo-immunotherapy (chemotherapy + immunotherapy) were continued.

ELIGIBILITY:
Inclusion Criteria:

-Patient's age: 18 years old - 80 years old -

* Rectal cancer patients diagnosed with adenocarcinoma by pathological examination of primary biopsy
* Patients with no prior treatment, preoperative clinical stage: cT3-4N+M0 rectal cancer patients (AJCC 8th);
* Patients who agree to undergo radical surgical treatment and have no contraindications to surgery as judged by the surgeon;
* No other multiple primary cancers;
* At least 1 measurable or evaluable lesion according to the efficacy evaluation criteria for solid tumors version 1.1 (RECIST v1.1);
* Expected survival time≥ 3 months;
* A score of 0-1 based on the United States Eastern Cooperative Oncology Group Performance Status Score (ECOG PS score);
* The investigator plans to give PD-1 monoclonal antibody combined with chemotherapy treatment regimen after evaluation, and signs informed consent.

Exclusion Criteria:

* Active, known or suspected autoimmune disease;
* Known history of primary immunodeficiency;
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
* Pregnant or lactating female patients;
* Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc., requiring emergency surgery;
* Uncontrolled intercurrent illness including but not limited to:
* People living with HIV (HIV antibody positive)
* Severe infections that are active or poorly clinically controlled
* Patients with active hepatitis
* Evidence of severe or uncontrolled systemic disease (e.g., severe psychiatric, neurological, epilepsy or dementia, unstable or incompensable respiratory, cardiovascular, hepatic or renal disease, uncontrolled hypertension [i.e., greater than or equal to CTCAE grade 2 hypertension despite medication]).
* Patients with active bleeding or new thrombotic disease, taking therapeutic dose of anticoagulant drugs or bleeding tendency, abnormal coagulation function (INR>1.5×ULN, APTT>1.5×ULN);
* Those who are currently undergoing clinical trials of other drugs;
* Other patients who are considered by the investigator to be unsuitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate（pCR） | assessment 2-4 weeks after surgery

SECONDARY OUTCOMES:
R0 resection rate | assessment 2-4 weeks after surgery
Disease-free survival at 3 years | from enrollment to three years after surgery
OS at 3 years | from enrollment to three years later
RECIST1.1 Objective response rate as assessed | 1-2 weeks before surgery
RECIST1.1 Disease control rate evaluated | 1-2 weeks before surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No